CLINICAL TRIAL: NCT01145300
Title: Relationship Between Exhaled Markers and Airway Pathology in Smokers With and Without Airflow Obstruction
Brief Title: Biomarkers in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Yvonne Nussbaumer-Ochsner, MD, Leiden University Medical Center
Other Study IDs: P10.045
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Inflammation; Small airways
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the leading causes of morbidity and mortality worldwide and is characterized by fixed airflow obstruction. The cornerstone of the disease is chronic inflammation leading to narrowing of the small airways and thus impairment of lung function. Compared to spirometry, the single breath N2-washout-test is more sensitive to identify the regional heterogeneity of bronchial airflow obstruction in the small airways.

The aim of this study is to evaluate whether there is a correlation between the sbN2-test, markers in exhaled air and the inflammatory cells in the small airways.

DETAILED DESCRIPTION:
The cornerstone of COPD is a chronic inflammation leading to narrowing of the small airways and thus impairment of lung function. Spirometry, the most frequently used pulmonary function test for diagnosing and monitoring disease, mostly reflects obstruction of the larger airways. The single breath N2-test, however, is more sensitive to identify the regional heterogeneity of bronchial airflow obstruction in the small airways, a main site of injury in COPD.

The aim of this study is to evaluate whether there is a correlation between the sbN2-test, markers in exhaled air and the inflammatory cells in the small airways.

This protocol describes a cross-sectional, explorative trial in at least 16 patients with COPD (up to GOLD III) and 8 patients without COPD who are scheduled for surgical resection for primary lung cancer. Immunohistological methods will be used to characterize the airways (large and small) inflammation pattern in macroscopically normal tissue containing small and large airways collected from sites distant from the tumor. Inflammatory markers will be measured in exhaled breath (exhaled breath condensate, exhaled NO) and be correlated to the sbN2 test. Breath patterns before and after lung cancer surgery will be assessed by the electronic nose and differential mobility spectrometry.

We hypothesize that the sbN2-test and inflammatory markers in exhaled breath reflect changes at peripheral tissue level. Therefore the results of the present study would lead to validation of these non-invasive tools for studies into the pathogenesis of obstructive lung disease, to increased knowledge about the relationship between airway inflammation and small airways obstruction, and may provide further support for the small airways as a specific target for inhaled drug delivery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject, age > 40 years, current or ex-smokers.
* Planned lung resection for primary lung cancer of any size.
* Patients with COPD: irreversible airflow limitation (postbronchodilator FEV1/FVC < 70% according to GOLD guidelines). Patients already receiving inhalative therapy can continue their medication. Patients showing a partial reversibility after bronchodilation (postbronchodilator FEV1 increase > 150 ml but < 200ml) and complaining respiratory symptoms (e.g. dyspnea at exertion) will be treated preoperatively with a short-acting beta-agonist to achieve optimal perioperative conditions.
* Patients without COPD: postbronchodilator FEV1/FVC > 70%.
* Patients have to be in clinical stable condition (no symptoms of respiratory tract infection for at least 2 weeks prior to the study).
* Written informed consent.

Exclusion Criteria:

* Patients with a history of asthma or other active lung disease.
* Lung resection for other reasons than lung cancer (e.g. infective diseases like bronchiectasis).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with and without COPD scheduled for lung resection for lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
1. Slope of the sbN2-test (phase III/IV) 2. Inflammatory markers in exhaled breath (NO, EBC, eNose, DMS) 3. Inflammation: localisation, numbers and profile of inflammatory cells in the large/small airways (neutrophils, macrophages, mastcells) | 1 week before surgery
  To demonstrate that the change in slope of the sbN2-test (phase III/IV) is correlated to an influx of inflammatory cells in the small airways (histology, morphology, immunopathology) and to inflammatory markers in exhaled breath in patients with normal and abnormal small airways function.

SECONDARY OUTCOMES:
Expression of the 1,25(OH)2D3 degrading enzyme CYP24A1 and antimicrobial peptides in small and large airways | within 1 week after surgery
  To assess whether there is a relationship between the expression of the 1,25(OH)2D3 degrading enzyme CYP24A1 and antimicrobial peptides in small and large airways in COPD patients and whether there is a correlation with local inflammation and lung function.
Markers in exhaled breath | 1 week before and 3 months after surgery
  To demonstrate that the presence of lung cancer per se is a condition leading to a change in the breath pattern. Exhaled breath patterns will be assessed by the eNose and the differential mobility spectrometry before and after lung cancer surgery.
Expression of macrophage markers (Mf1 and Mf2) and chymase/tryptase in mast cell subsets | within 1 week after surgery
  To assess whether there is a difference in expression of macrophage Mf1 and Mf2 markers, and in mast cell subsets (chymase/tryptase positive vs. tryptase positive) in small and large airways from patients with COPD at lung tissue level.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus F. Rabe, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Department of Pulmonology, Leiden University Medical Center, Leiden, Netherlands